CLINICAL TRIAL: NCT06625125
Title: The Differential Effects of Mindfulness-Based Intervention and Progressive Muscle Relaxation on Expression Suppression, Cognitive Reappraisal, and Perceived Stress in Patients With End-Stage Renal Disease: A Randomized Trial
Brief Title: PMR vs MM for Patients on Hemodialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hossam Najjem Alhawatmeh, Associate professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/369
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; End stage renal disease; Mindfulness meditation; Progressive muscle relaxation; Cognitive reappraisal; Behavioral suppression; Perceived stress
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the participants' random assignment to either the experimental or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with ESRD receiving mindfulness-based intervention (Experimental): The mindful mediators are asked to act as neutral observers who quietly attend to, notice, and let go of internal and external stimuli (present experiences) such as thoughts, feelings, physical sensations, and sounds without reactions, evaluation, and judgments. (Smith, 2005).
  The subjects in the mindfulness-based intervention (MBI) group will receive 30 minutes individually administered, guided, chairside interventions during their hemodialysis sessions, three times a week over eight weeks (Alhawatmeh et al., 2022; Thomas et al., 2017). Subjects in this group will receive their assigned intervention developed by the principal investigator (PI) according to the Smith's MBI protocol that will provide intervention instructions. During the eight weeks and at bedtime at night, the subjects will be optionally encouraged to practice the intervention at home.
  Interventions: Behavioral: Mindfulness-based intervention
- Patients with ESRD receiving progressive muscle relaxation (Active Comparator): The progressive muscle relaxation (PMR) group will receive the ABC version of PMR (Smith, 2005). This abbreviated version of PMR involves a tense-let go exercise of 11 muscle groups including hand, arm, arm and sides, back, shoulder, face, front of neck, stomach, chest, leg, and foot.
  As the MBI group, the subjects in the PMR group will receive 30 minutes individually administered, guided, chairside interventions during their hemodialysis sessions, three times a week over eight weeks. Subjects in this group will receive their assigned intervention developed by the principal investigator (PI) according to the Smith's PMR protocol that will provide intervention instructions. During the eight weeks and at bedtime at night, the subjects will be optionally encouraged to practice the intervention at home.
  Interventions: Behavioral: Progressive muscle relaxation
- Patients with ESRD receiving the hospital traditional care (No Intervention): The control group will not receive any intervention from the study researchers

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — The mindful mediators are asked to act as neutral observers who quietly attend to, notice, and let go of internal and external stimuli (present experiences) such as thoughts, feelings, physical sensations, and sounds without reactions, evaluation, and judgments. (Smith, 2005).
  The subjects in the mindfulness-based intervention (MBI) group will receive 30 minutes individually administered, guided, chairside interventions during their hemodialysis sessions, three times a week over eight weeks (Alhawatmeh et al., 2022; Thomas et al., 2017). Subjects in this group will receive their assigned intervention developed by the principal investigator (PI) according to the Smith's MBI protocol that will provide intervention instructions. During the eight weeks and at bedtime at night, the subjects will be optionally encouraged to practice the intervention at home.
  Arms: Patients with ESRD receiving mindfulness-based intervention
Behavioral: Progressive muscle relaxation — he progressive muscle relaxation (PMR) group will receive the ABC version of PMR (Smith, 2005). This abbreviated version of PMR involves a tense-let go exercise of 11 muscle groups including hand, arm, arm and sides, back, shoulder, face, front of neck, stomach, chest, leg, and foot.
  As the MBI group, the subjects in the PMR group will receive 30 minutes individually administered, guided, chairside interventions during their hemodialysis sessions, three times a week over eight weeks. Subjects in this group will receive their assigned intervention developed by the principal investigator (PI) according to the Smith's PMR protocol that will provide intervention instructions. During the eight weeks and at bedtime at night, the subjects will be optionally encouraged to practice the intervention at home.
  Arms: Patients with ESRD receiving progressive muscle relaxation

SUMMARY:
Background: Hemodialysis is considered as an effective therapy to remove harmful waste from the body and to improve the quality of life in patients suffering from end-stage renal disease (ESRD). However, patients who receive hemodialysis perceive various stressors that are harmful to their physical and psychological well-being. Therefore, it is necessary to implement effective and practical therapeutic strategies to enhance the quality of life in this population. Mindfulness-based intervention (MBI) and progressive muscle relaxation (PMR) are effective mind-body connection programs that are inadequately used in patients undergoing hemodialysis.

Objectives: This study will examine the differential effects of mindfulness-based intervention (MBI) and progressive muscle relaxation (PMR) on expression suppression, cognitive reappraisal, and perceived Stress in Patients with End-Stage Renal Disease undergoing hemodialysis in Jordan.

Methods: An experimental parallel control, randomized design will be implemented among 159 PwESRD undergoing hemodialysis in a big referral Hospital in Jordan. Simple random assignation will be used to create three equal groups including PMR, MBI, and control groups (N= each). Both groups will practice their assigned intervention over five weeks (with three half-hour sessions per week) during hemodialysis sessions. The study variables will be measured for the three groups at the outset and eight weeks after initiation. Variables will be measured by the self-reporting questionnaire including sociodemographic characteristic sheet, the Mindfulness attention awareness scale (MAAS) the Perceived Stress Scale (PSS), and the Emotion Regulation Questionnaire (ERQ). Repeated measures analysis of variance (RM ANOVA) will be used to analyze the main study data.

DETAILED DESCRIPTION:
Background

End-stage renal disease (ESRD) is a serious health issue that affects 10-14% of the adult population worldwide. ESRD, which has become one of the top causes of death on a global scale, is characterized by the kidneys only operating at 10 to 15% of their normal capacity. In Jordan, according to its registry of renal patients, the Ministry of Health (MoH) reported 7747 of such patients by the beginning of 2021, comprising 7290 Jordanian nationals (94.1%), and 457 (5.9%) non-Jordanians.

Hemodialysis (HD) is a vitally important treatment for patients with ESRD (PwESRD), that extends life by excreting the body's toxic metabolic waste. However, the difficulties that patients on HD confront are various and significant, putting such patients under sever level of perceived stress. HD is one of the most stressful treatments because it has so many stressors, including the requirement to visit medical facilities, to stay a significant amount of time there, to take prescribed medications, to manage diet and fluid intake, and to seriously alter lifestyle choices and possibilities. Although acute stress works to maintain bodily hemostasis, repeated exposures to stress over time can negatively affect patients' physical, psychological and social health, jeopardizing their quality of life.

Globally, the use of complementary and alternative medicine (CAM) has grown over the past 20 years. Mind-body interventions are a core part of CAM. Mind body interventions is described by the National Center for Complementary and Integrative Health as a collection of practices or techniques that primarily concentrate on the relationships between the mind, body, and behavior and how those relationships affect one's stress and quality of life. It includes practices like music therapy, yoga, hypnosis, meditation including mindfulness, and relaxation. Mindfulness-based intervention (MBI) and progressive muscle relaxation (PMR) are the most well-established and widely used complementary therapies.

MBI is defined as moment-by-moment awareness of daily experiences with the attitudes of acceptance and non-judgment. PMR is defined as the act of regular and systematic tensing and relaxing different muscle groups with focused attention on relaxation and tension of these muscles. These Mind-body therapies, recently increasing their popularity in Jordan, are easily accessible, easy to learn and inexpensive. Mind-body interventions were classified as focused attention practice and open monitoring practice, which have differential treatment mechanisms and effects. Focused attention practices involve sustaining attention to a single stimulus such as tension and relaxation of muscles. However, open monitoring practices involve a receptive awareness or monitoring of all stimuli that arise moment-to-moment. Accordingly, MBI can be classified as an open monitoring (OM) practice while PMR classified as a focused attention (FA) practice.

There have been studies supporting the potential positive effects of MBI and PMR on perceived stress among patients undergoing hemodialysis. However, the mechanisms of the beneficial effects of both therapies such as MBI and PMR on perceived stress among such patients have been rarely studied. In recent years, there has been an increasing interest in identifying the underlying mechanisms of mind body therapies because of growing evidence of its benefits on mental disorders and physical well-being. A number of theoretical approaches have been suggested to identify how MBI or PMR affects perceived stress. It has been proposed that the mechanisms of open monitoring practice such as MBI potentially involve changes in emotion regulation strategies such as stress reappraisal. However, focused attention practice such as PMR can affect health through increased expression suppression as an emotional regulation strategy.

Reappraisal is an emotional regulation strategy that reduces emotional responses through a change of the meaning of a certain stressful situation. Thus, it has a long-term effect on perceived stress. Expressive suppression, However, is an emotional regulation strategy that inhibits behaviors related to emotional responses (e.g., facial expressions) and decrease the emotions' expression, not their experience. Notably, reappraisal has been emphasized as one of the mechanisms through which MBI works. However, expression may be one of the mechanisms through which PMR works. Expressive suppression opposes important aspect of mindfulness, described as the awareness and acceptance of emotions, but matches with the avoidance coping, which has lower effect on perceived stress and its effects on stress are short-lived. Accordingly, mindfulness has been reported to be positively related to cognitive reappraisal and negatively with expressive suppression.

It is explained that psychosomatic health problems such as perceived stress result from the conditioned automatic cycle of association formed from distressing thoughts and associated feelings and sensations that is initiated when attention is not consciously or intentionally directed. For example, when one experiences a certain threat (alarming thought), emotion (e.g. fair) is evoked that is accompanied by physical sensations (e. g. muscle tension). Our habitual reactions to feelings or sensations are to pursue those that are evaluated as pleasant and to avoid those that are evaluated unpleasant. These habitual reactions are expressed as mental events or thoughts that rapidly follow the initial alarming thought, feeling and sensation. The mental events or thoughts that follow the initial thought, feeling, and sensation also have associated feelings and sensations. This associational cycle is maintained as long as attention remains preoccupied with or embedded in these components in an unconscious way that, in turn, leads to chronically elevated psychosomatic stress responses. In OM meditation, practitioner who intentionally pays attention to sensations, emotions, and thoughts moment- to- moment will become aware of that these experiences are transitory that arise and pass away and do not constitute lasing entity and there is no need take steps to avoid them. The effect of this state of nonreactive awareness on stress responses is mediated by the emotional regulation strategy of cognitive reappraisal. Cognitive reappraisal is defined as re-evaluating the meaning of a distressed stimulus to change the negative emotional responses. In short, being aware of that the emotions, sensations and thoughts are transitory, and not-lasting objects that arise and pass away cultivate the belief that these experiences are passing events that does not endanger health if people do not habitually avoid or be over-engaged with them (cognitive reappraisal).

FA practice such as PMR can lead to positive outcomes related to psychosomatic health, however, it works through mechanisms that are different from the mechanisms employed in OM meditation. The effect of FA meditation on stress responses is mediated by the emotion regulation strategy of thought suppression, not cognitive reappraisal as Lutz et al. explained. Expressive suppression is defined as intentionally removing a distress thought or behavior from conscious awareness. Attentional resources are limited, which means that attention can be paid to only one object at a time. Thus, if attention is sufficiently sustained on an object such as sensations of breath or muscular tension and relaxation, this prevents practitioner to remain preoccupied with or aware of other objects in that moment such as distressed thoughts and in turn decrease stress responses. FA meditation does not lead to cognitive reappraisal. In FA meditation, practitioner tries to not evaluate or be judgmental about the distractor (stimulus) and in turn creates a temporary state of "non-appraisal", not reappraisal. This state of non-appraisal resulting from the inhibition thought, or behaviors is temporary that ends when attention lapses from the meditation object (e.g. muscle tension and relaxation), unlike the cognitive reappraisal evoked by OM meditation, which have long-lasting effect on perceived stress.

To the best of our knowledge, however, these theoretical approaches that explain the differential mechanism and effect of open monitoring practice (e.g. MBI) and focused attention practice (e.g. PMR) on perceived stress have been rarely empirically supported., especially in patients with ESRD. Thus, the purpose of this study is to compare the differential effects of MBI and PMR on cognitive reappraisal, expressive suppression, and perceived stress in patients with ESRD undergoing hemodialysis.

Methods

Design and Setting

An experimental study with a randomized, repeated-measures, parallel control design will be conducted in hemodialysis units in two Jordanian hospitals- King Abdullah University Hospital and the Prince Rashid Military Hospital.

Participants

The G*Power (3.1 software's) analysis suggested that a sample size of 159 participants will be adequate to study as per an analysis of variance (ANOVA), given a Cronbach's alpha (α) level of significance of .05, a power level of 0.8, and a moderate effect size of 0.25.

Interventions

The MBI and PMR groups will receive MBI and PMR respectively according to Smith's (2005) protocols. It is standardized theory-based interventions found to be effective in improving physical and psychological health outcomes. The subjects in both groups will receive 30 minutes individually administered, guided, chairside interventions during their hemodialysis sessions, three times a week over eight weeks (e.g. PMR group will receive PMR protocol, but MBI will receive MBI protocol). This approach has been used and found to be feasible and effective for patients receiving hemodialysis. Subjects in both groups will receive audio recording of their assigned intervention developed by the principal investigator (PI) according to the Smith's MBI protocol that will provide intervention instructions. The assigned audio recording will be sent to the subjects via WhatsApp (iOS and Android) to be used during the intervention sessions, to warrant the consistent delivery of the intervention. To ensure that they can practice effectively, they will be supervised by a study researcher during the intervention sessions. During the eight weeks and at bedtime at night, the subjects will be optionally encouraged to practice the intervention at home.

Before the beginning of the self-administered intervention sessions, face-to face foundation Course (2 hours) will be conducted by the certified study researcher who educated and trained the subjects on their assigned interventions in separate rooms about the basics and protocol of their intervention. The certified study researcher who had an advanced degree in nursing and 12 years of nursing experience received an extensive training workshop on "Mind-Body Practice". A checklist will be developed and maintained by the PI including all steps of the intervention (each step and the length of time to spend on each step) to achieve high degrees of adherence. The subjects were requested not to take any psychotherapies or psychopharmacological medications if they are necessarily needed, and to notify the PI of such treatments were taken during the intervention. Patients' medical records were checked regularly during the intervention to warrant they did not receive any psychological and analgesic medication. Any potential interruption (e.g., the dialysis machine alarm) was handled instantly by the attending nurses.

MBI

The mindful mediators are asked to act as neutral observers who quietly attend to, notice, and let go of internal and external stimuli (present experiences) such as thoughts, feelings, physical sensations, and sounds without reactions, evaluation, and judgments. They are asked not to make any attempts to think about or push away these stimuli. They easily allow each stimulus that enter awareness come and go and wait for the subsequent stimuli. They should not be concerned about distractions. Whenever they are distracted, they observe and label and let them go as yet other passing stimuli (Ah, a distraction… how interesting").

PMR

The PMR group will receive the ABC version of PMR. This abbreviated version of APMR involves a tense-let go exercise of 11 muscle groups including hand, arm, arm and sides, back, shoulder, face, front of neck, stomach, chest, leg, and foot. This tense-let go exercise is performed twice for each muscle group. The tensing up phase for each muscle group should last for 5 to 10 seconds and the letting go phase for 20-30 seconds. Simultaneously, the subjects are asked to pay attention to the sensations of muscle tension and relaxation. After the tense-let go exercise, subjects are asked to systematically scan the muscle groups to notice and let go any remaining muscle tension. The entire exercise should take around 30 minutes, not counting instructions and times of measurement.

Control Group: they will receive traditional care used in the hospital.

Intervention fidelity

To achieve high levels of adherence, a checklist involving all steps of both interventions will be maintained (see Appendix G). The certified study researcher will have a hard copy checklist to refer to, which includes each step and the length of time to spend on each step. The development of these checklists will be based on Smith's protocols. Delivery of interventions will be immediately evaluated by the certified study researcher using the checklists after each training session.

Procedure

First, permission to use the study instruments will be sought. The researchers will carry out the participant recruitment after receiving permission from the hospital officials to conduct the study. The patients will be contacted by a study researcher who will provide a thorough explanation of the study's goals and protocol. Patients who will complete the eligibility requirements and agree to participate in the study will be asked to sign a consent form. A simple computer-generated sequence will then be used for random assignment of participants into the study groups, each of which had 53 participants (total N = 159). A study researcher who has a doctoral degree in nursing will implement the randomization. This study researcher will not be involved in other parts of the study. After that, the baseline measurements for all study outcomes using the study instruments and demographic characteristics will be completed by the participants, utilizing the self-report questionnaires (T0) for the study variables.

The PMR and MBI groups will receive the Smith Protocols of PMR and MBI respectively. This will be administered to the group participants individually during their normal HD sessions, over the course of half an hour per session. The Protocol will be demonstrated to be practical and efficacious for patients on HD. Smith (2005) based the Protocol on the "ABC Relaxation Theory", and advised their delivery via 2-5 half-hour sessions per week. Such MBI and PMR are intended to induce a state of calm, without stress, and to subsequently contribute to improved health and wellbeing. For particular application among patients undergoing HD, 400 total minutes of mind-body intervention delivery is expected to be necessary to achieve substantive benefits. With this in mind, the study groups' participants in this study will receive three half-hour sessions per week over five weeks, collectively totaling 450 minutes. Additionally, the study groups' participants will also be delivered a two-hour Foundation Course before initiating the actual training sessions. This course will communicate to participants the fundamentals, intended outcomes, and procedures of the interventions.

To give the assigned intervention to patients, a research assistant with a BSc in nursing, 15 years of nursing experience, a diploma in nephrology, a master's in psychology will be asked; however, she will be excluded from the procedure of recruiting participants, as well as the data collection and randomization steps. This researcher assistant had extensive training in Mind body therapies. Participants' confidentiality and privacy will be ensured at all stages of this study, and curtains will be closed to give each participant total privacy during the intervention delivery. Additionally, the participants themselves in both study group will be requested not to communicate the details of the intervention with anybody during the study.

The study variables (Mindfulness trait, perceived stress, expression suppression, and cognitive reappraisal) will be measured for three groups at the outset, and 8 weeks after initiation to detect improvements in the study outcomes over time. An well-trained research assistant with a master's in nursing, who will be unaware of the randomization and allocation steps, will undertake measurement of the study variables at both time points, within conditions of privacy at the dialysis facility.

Ethical Considerations

Jordan University of Science and Technology's Institutional Review Board (IRB) will approve the proposed study. Participants who agree to participate in the study will be asked to sign a written consent form that explains the purpose and scope of the research. They will be confirmed that they will have the freedom to reject participation in the study and that such rejection will not affect the care they receive. They will be assured that the research data will be stored in a secure location in a locked cabinet, with numbers replacing their names to avoid their identification. No patients will be excluded from the trial because of their gender, race, or nationality. During the intervention, if any patient felt dizzy or uncomfortable, the intervention will be stopped, and the doctor will be informed immediately.

Data Analyses

SPSS (version 23) will be used to statistically analyze the results, with descriptive statistics and measurement level-appropriate dispersion and central tendency measures for the variables and sample. For example, means and SD were calculated for the dependent variables that were measured on interval level of measurement, and frequency were calculated for the categorical variables such as gender. Initial analyses will be undertaken to be certain of successful covariate randomization and statistical test assumptions. One-way ANOVA will be used to test the significant differences in trait mindfulness, perceived stress, expression suppression and cognitive reappraisal between the study groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with ESRD undergoing hemodialysis at least three sessions a week
* being at least 18 years old
* having a smartphone
* being capable of reading and writing in Arabic

Exclusion Criteria:

* Patients under psychotherapy or taking regular psychopharmacological and analgesic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | From enrollment to the end of treatment at 8 weeks
  An Arabic version of the Perceived Stress Scale (PSS) was used to measure the degree to which situations in one's life are appraised as stressful (unpredictable, uncontrollable, and overloaded) (Almadi, et al., 2012). It includes 10 items measured on a 5-point Likert scale (0=never, 4= very often), which are relatively free of content specific to any subpopulation group. The scores range from 0 to 40 with higher score indicating higher levels of perceived stress (stressful appraisal) (Cohen, et al., 1983). PSS has been validated for use with college students. Internal consistency coefficients for the PSS ranged from .84 to 36, and test- retest reliability is .85 (Cohen et al., 1983). The Arabic Perceived Stress Scale showed adequate reliability and validity and considered a suitable instrument to assess perceived stress in Arabic people (Almadi et al., 2012).
Emotion Regulation Questionnaire (ERQ) | From enrollment to the end of treatment at 8 weeks
  An Arabic version of ERQ will be used to measure emotion regulation abilities including cognitive reappraisal and expression suppression. The questionnaire is a 7-point Likert-type scale, with two subscales including cognitive reappraisal (6 items) and expressive suppression (4 items). The scale items are rated on a scale from 1 (strongly disagree) to 7 (strongly agree). The higher scores indicate greater emotion regulation abilities such as cognitive reappraisal and expressive suppression (Gross & John, 2003). Arabic version showed valid and reliable results among Arabic Gulf population and Jordanian patients with ESRD (Alhawatmeh et al. 2022; Keshky, 2018).

SECONDARY OUTCOMES:
The Mindful Attention Awareness Scale (MAAS) | From enrollment to the end of treatment at 8 weeks
  The MAAS is a widely used self-report measure designed to assess an individual's trait mindfulness-their general capacity to be present and attentive to ongoing experiences in daily life. The MAAS typically consists of 15 items. Patients rate how frequently they experience various characteristics of mindfulness in day-to-day activities. Participants rate each item on a Likert-type scale. This scale indicates frequency of experiences from "1: almost always" to "5: almost never" (Brown & Ryan, 2003). The total Score on the MAAS range from 15 to 75, with ahigher scores indicating higher levels of trait mindfulness. The scale has been applied extensively in clinical and scientific contexts. It investigates connections between many facets of mental health and wellbeing and mindfulness (Brown & Ryan, 2003). Strong convergent validity and internal consistency are demonstrated by Arabic MAAS among Arab hemodialysis patients (Alhawatmeh et al., 2022).

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Alhawatmeh, Principal Investigator — Hossam alhawatmeh, assistant professor, Jordan university of science and technology
Locations (1):
- Prince Rashid Military Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
The data is not available to other researchers due to ethical restrictions

REFERENCES:
- [Background] Alhawatmeh H, Alshammari S, Rababah JA. Effects of mindfulness meditation on trait mindfulness, perceived stress, emotion regulation, and quality of life in hemodialysis patients: A randomized controlled trial. Int J Nurs Sci. 2022 Mar 8;9(2):139-146. doi: 10.1016/j.ijnss.2022.03.004. eCollection 2022 Apr. PMID 35509694
- [Background] Almadi T, Cathers I, Hamdan Mansour AM, Chow CM. An Arabic version of the perceived stress scale: translation and validation study. Int J Nurs Stud. 2012 Jan;49(1):84-9. doi: 10.1016/j.ijnurstu.2011.07.012. Epub 2011 Aug 17. PMID 21851941
- [Background] Beevers, C. G., Wenzlaff, R. M., Hayes, A. M., & Scott, W. D. (1999). Depression and the ironic effects of thought suppression: Therapeutic strategies for improving mental control. Clinical Psychology: Science and Practice, 6,133-148
- [Background] Bennett PN, Ngo T, Kalife C, Schiller B. Improving wellbeing in patients undergoing dialysis: Can meditation help? Semin Dial. 2018 Jan;31(1):59-64. doi: 10.1111/sdi.12656. Epub 2017 Nov 2. PMID 29098724
- [Background] Carmody, J. (2009). Evolving conceptions of mindfulness in clinical settings. Journal of Cognitive Psychotherapy, 23, 270-280.
- [Background] Chambers R, Gullone E, Allen NB. Mindful emotion regulation: An integrative review. Clin Psychol Rev. 2009 Aug;29(6):560-72. doi: 10.1016/j.cpr.2009.06.005. Epub 2009 Jun 23. PMID 19632752
- [Background] Chu SWF, Yeam CT, Low LL, Tay WY, Foo WYM, Seng JJB. The role of mind-body interventions in pre-dialysis chronic kidney disease and dialysis patients - A systematic review of literature. Complement Ther Med. 2021 Mar;57:102652. doi: 10.1016/j.ctim.2020.102652. Epub 2020 Dec 26. PMID 33373760
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Dehghan M, Namjoo Z, Bahrami A, Tajedini H, Shamsaddini-Lori Z, Zarei A, Dehghani M, Ranjbar MS, Rafiee Sarbijan Nasab F. The use of complementary and alternative medicines, and quality of life in patients under hemodialysis: A survey in southeast Iran. Complement Ther Med. 2020 Jun;51:102431. doi: 10.1016/j.ctim.2020.102431. Epub 2020 May 21. PMID 32507442
- [Background] Holzel BK, Lazar SW, Gard T, Schuman-Olivier Z, Vago DR, Ott U. How Does Mindfulness Meditation Work? Proposing Mechanisms of Action From a Conceptual and Neural Perspective. Perspect Psychol Sci. 2011 Nov;6(6):537-59. doi: 10.1177/1745691611419671. PMID 26168376
- [Background] Garland EL, Roberts RL, Hanley AW, Zeidan F, Keefe FJ. The Mindful Reappraisal of Pain Scale (MRPS): Validation of a New Measure of Psychological Mechanisms of Mindfulness-Based Analgesia. Mindfulness (N Y). 2023 Jan;14(1):192-204. doi: 10.1007/s12671-022-02034-y. Epub 2022 Dec 16. PMID 37901118
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Keshky, M. E. E. (2018). Keshky ME. Factor Structure, Reliability and Validity of the Arabic Version of the Emotion Regulation Questionnaire (ERQ) in a Sample of Saudi Children and Adolescents. International Journal of Psychology and Behavioral Sciences. 2018;8(2):22-30.
- [Background] Kabat-Zinn, J. (1990). Full catastrophe living: Using the wisdom of your body and mind to face stress, pain, and illness. PsycCRITIQUES, 37(6), 609-609. https://doi.org/10.1037/032287
- [Background] Lutz A, Slagter HA, Dunne JD, Davidson RJ. Attention regulation and monitoring in meditation. Trends Cogn Sci. 2008 Apr;12(4):163-9. doi: 10.1016/j.tics.2008.01.005. Epub 2008 Mar 10. PMID 18329323
- [Background] Nassim M, Park H, Dikaios E, Potes A, Elbaz S, Mc Veigh C, Lipman M, Novak M, Trinh E, Alam A, Suri RS, Thomas Z, Torres-Platas S, Vasudev A, Sasi N, Gautier M, Mucsi I, Noble H, Rej S. Brief Mindfulness Intervention vs. Health Enhancement Program for Patients Undergoing Dialysis: A Randomized Controlled Trial. Healthcare (Basel). 2021 Jun 1;9(6):659. doi: 10.3390/healthcare9060659. PMID 34205915
- [Background] Parmentier FBR, Garcia-Toro M, Garcia-Campayo J, Yanez AM, Andres P, Gili M. Mindfulness and Symptoms of Depression and Anxiety in the General Population: The Mediating Roles of Worry, Rumination, Reappraisal and Suppression. Front Psychol. 2019 Mar 8;10:506. doi: 10.3389/fpsyg.2019.00506. eCollection 2019. PMID 30906276
- [Background] Ray RD, McRae K, Ochsner KN, Gross JJ. Cognitive reappraisal of negative affect: converging evidence from EMG and self-report. Emotion. 2010 Aug;10(4):587-92. doi: 10.1037/a0019015. PMID 20677875
- [Background] Saleh, W., Maani, N., & Sharkas, G. (2020). The Hashemite Kingdom of Jordan Ministry of Health 13th annual report. Ministry of Health.
- [Background] Smith, J. C. (2005). Relaxation, meditation, & mindfulness: A mental health practitioner's guide to new and traditional approaches. Springer Publishing Company.
- [Background] Thomas Z, Novak M, Platas SGT, Gautier M, Holgin AP, Fox R, Segal M, Looper KJ, Lipman M, Selchen S, Mucsi I, Herrmann N, Rej S. Brief Mindfulness Meditation for Depression and Anxiety Symptoms in Patients Undergoing Hemodialysis: A Pilot Feasibility Study. Clin J Am Soc Nephrol. 2017 Dec 7;12(12):2008-2015. doi: 10.2215/CJN.03900417. Epub 2017 Oct 12. PMID 29025788
- [Background] Travis F, Shear J. Focused attention, open monitoring and automatic self-transcending: Categories to organize meditations from Vedic, Buddhist and Chinese traditions. Conscious Cogn. 2010 Dec;19(4):1110-8. doi: 10.1016/j.concog.2010.01.007. Epub 2010 Feb 18. PMID 20167507
- [Background] Zhang D, Lee EKP, Mak ECW, Ho CY, Wong SYS. Mindfulness-based interventions: an overall review. Br Med Bull. 2021 Jun 10;138(1):41-57. doi: 10.1093/bmb/ldab005. PMID 33884400
- [Background] Wenzlaff RM, Wegner DM. Thought suppression. Annu Rev Psychol. 2000;51:59-91. doi: 10.1146/annurev.psych.51.1.59. PMID 10751965